CLINICAL TRIAL: NCT04485286
Title: Evaluation of PET Probe [68Ga]CBP8 in the Detection of Radiation Induced Tissue Injury
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter Caravan, Professor of Radiology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020P001899; R44CA250771 (NIH); K08CA259626 (NIH)
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer; Radiation Fibrosis; Radiation Induced Lung Injury; Pancreas Cancer
Keywords: fibrosis; positron emission tomography
MeSH Terms: conditions — Lung Neoplasms; Radiation Fibrosis Syndrome; Pancreatic Neoplasms; Fibrosis

STUDY DESIGN:
Intervention Model Description: Eligible subjects planning on receiving radiation for lung cancer or pancreatic cancer will be enrolled to undergo imaging with the PET Probe [68Ga]CBP8.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lung Cancer or Pancreatic Cancer Subjects Undergoing Radiation Therapy (Experimental): Lung cancer or pancreatic cancer patients will receive [68Ga]CBP8 and undergo PET imaging 1) prior to radiation therapy and 2) 3-6 months after radiation therapy
  Interventions: Drug: [68Ga]CBP8

INTERVENTIONS:
Drug: [68Ga]CBP8 — Up to 15 mCi of [68Ga]CBP8 will be administered to each subject. Each subject will undergo baseline imaging prior to radiation and again 3-6 months after radiation therapy.

SUMMARY:
The goal of this study is to investigate the efficacy of [68Ga]CBP8 to detect collagen deposition in radiation induced tissue injury.

DETAILED DESCRIPTION:
Detailed Description:

The investigators have developed [68Ga]CBP8, a gallium-68 labeled collagen binding PET imaging probe, which selectively binds collagen type I. Collagen deposition is a pivotal event in several human conditions including radiation induced lung injury and in response to radiation therapy in pancreatic cancer. The investigator's studies in murine models of lung injury including radiation induced lung injury showed that [68Ga]CBP8 binds collagen with high affinity and has excellent pharmacological and pharmacokinetic profiles with high target uptake and low retention in background tissues and organs. [68Ga]CBP8 was shown in a mouse model to be effective for detecting lung fibrosis. [68Ga]CBP8 showed high specificity for pulmonary fibrosis and high target:background ratios in diseased animals. In addition, [68Ga]CBP8 could be used to monitor response to treatment. Ex vivo analysis of lung tissue from patients with idiopathic pulmonary fibrosis (IPF) supported the animal findings.

The investigators have conducted preliminary studies in humans with IPF and demonstrated a significant increase in [68Ga]CBP8 signal in subjects with IPF vs healthy controls.

The investigators thus aim to evaluate [68Ga]CBP8 in human subjects with radiation induced lung injury and in patients undergoing radiation therapy for pancreatic cancer:

To establish the ability of [68Ga]CBP8-PET to detect radiation-induced fibrosis in lung or pancreatic cancer patients through the course of disease development with repeated measures, and correlate signal with standard measures of radiation induced tissue injury such as HRCT or MRI.

ELIGIBILITY:
Inclusion Criteria for lung cancer subjects:

* Eligible patients will be those harboring locally advanced clinical stage I-III NSCLC who are not eligible for surgical resection, or those with stage IIIa NSCLC who are deemed candidates for multi-modality therapy, i.e. concurrent chemotherapy and radiation followed by pulmonary resection.
* Age greater than 18 years
* Have the ability to give written informed consent.
* No tobacco use within the prior 6 months.

Inclusion Criteria for pancreatic cancer subjects:

* Age ≥ 18 years.
* Life expectancy of greater than 3 months.
* Ability to understand and the willingness to sign a written informed consent document.
* Histologically or cytologically confirmed diagnosis of PDAC.
* Tumor should be confirmed with imaging based on the standard-of-care baseline abdominal CT performed within 1 month before study visit 1.
* Core samples for initial diagnosis must be available at the Department of Pathology at Massachusetts General Hospital.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational imaging and standard treatment regimen are eligible for this trial.
* Scheduled study visit 1 within 1 month prior to starting neoadjuvant chemoradiotherapy (CRT)
* Subjects undergo neoadjuvant chemotherapy followed by radiotherapy (CRT) as part of their standard clinical care and based on institutional standards.
* Scheduled surgical pancreas resection within 1 month after post-CRT study visit.
* Subjects are required to undergo pre-surgical CT of abdomen within 1 month after completion of standard neoadjuvant CRT as part of routine clinical work-up.

Exclusion Criteria for lung cancer subjects:

* Electrical implants such as cardiac pacemaker or perfusion pump
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, or steel implants ferromagnetic objects such as jewelry or metal clips in clothing;
* Pregnant or breastfeeding (a negative quantitative serum hCG pregnancy test is required for females having child-bearing potential before the subject can participate);
* Claustrophobic reactions;
* Research-related radiation exposure exceeds current Radiology Department guidelines (i.e. 50 mSv in the prior 12 months);
* Unable to lie comfortably on a bed inside the MR-PET;
* Body weight of > 300 lbs (weight limit of the MRI table);
* Determined by the investigator(s) to be clinically unsuitable for the study (e.g. based on screening visit and/or during study procedures);
* Known history of pulmonary disease (Except lung cancer or smoking related lung disease,)
* Pneumonia or other acute respiratory illness within 6 weeks of study entry, pneumonia defined with elevated WBC, fever, infiltrate on CXR and need for antibiotics

Exclusion Criteria for pancreatic cancer subjects:

* History of radiotherapy to the upper abdomen in the past.
* History of reaction to MRI contrast (Gadoterate meglumine)
* Clinical or imaging diagnosis of acute pancreatitis within 6 weeks prior to study visit
* Participants with uncontrolled intercurrent illness or if determined by the investigator(s) to be clinically unsuitable for the study (e.g. based on screening and/or during study).
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Electrical implants such as cardiac pacemaker or perfusion pump;
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, or steel implants ferromagnetic objects such as jewelry or metal clips in clothing;
* eGFR of less than 30 mL/min/1.73 m2 within the past 90 days;
* Pregnant or breastfeeding (a negative quantitative serum hCG pregnancy test is required for females having child-bearing potential at each PET/MRI study visit;
* Claustrophobic reactions;
* Research-related radiation exposure exceeds current Radiology Department guidelines (i.e. 50 mSv in the prior 12 months);
* Unable to lie comfortably on a bed inside the MR-PET;
* BMI > 33 (limit of the PET-MRI table)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-07-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Ability of [68Ga]CBP8 to detect collagen deposition in areas of radiation injury. | 3-6 Months
  Probe uptake will be measured in lung cancer or pancreatic cancer patients 1) prior to radiation therapy and 2) 3-6 months after radiation therapy. We expect [68Ga]CBP8 signal to be increased in post radiation measurements over pre-radiation measurements in areas of irradiated tissue. Furthermore we expect that these areas will go on to develop radiation fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lanuti, MD, Principal Investigator — Massachusetts General Hospital; Shadi Esfahani, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montesi SB, Izquierdo-Garcia D, Desogere P, Abston E, Liang LL, Digumarthy S, Seethamraju R, Lanuti M, Caravan P, Catana C. Type I Collagen-targeted Positron Emission Tomography Imaging in Idiopathic Pulmonary Fibrosis: First-in-Human Studies. Am J Respir Crit Care Med. 2019 Jul 15;200(2):258-261. doi: 10.1164/rccm.201903-0503LE. No abstract available. PMID 31161770
- [Background] Desogere P, Tapias LF, Rietz TA, Rotile N, Blasi F, Day H, Elliott J, Fuchs BC, Lanuti M, Caravan P. Optimization of a Collagen-Targeted PET Probe for Molecular Imaging of Pulmonary Fibrosis. J Nucl Med. 2017 Dec;58(12):1991-1996. doi: 10.2967/jnumed.117.193532. Epub 2017 Jun 13. PMID 28611243
- [Background] Desogere P, Tapias LF, Hariri LP, Rotile NJ, Rietz TA, Probst CK, Blasi F, Day H, Mino-Kenudson M, Weinreb P, Violette SM, Fuchs BC, Tager AM, Lanuti M, Caravan P. Type I collagen-targeted PET probe for pulmonary fibrosis detection and staging in preclinical models. Sci Transl Med. 2017 Apr 5;9(384):eaaf4696. doi: 10.1126/scitranslmed.aaf4696. PMID 28381537
- [Derived] Abston E, Zhou IY, Saenger JA, Shuvaev S, Akam E, Esfahani SA, Hariri LP, Rotile NJ, Crowley E, Montesi SB, Humblet V, Arabasz G, Catana C, Fintelmann FJ, Caravan P, Lanuti M. Noninvasive Quantification of Radiation-Induced Lung Injury using a Targeted Molecular Imaging Probe. medRxiv [Preprint]. 2023 Sep 26:2023.09.25.23295897. doi: 10.1101/2023.09.25.23295897. PMID 37808864